CLINICAL TRIAL: NCT02952209
Title: The Effect of Alveolar Ridge Preservation After Tooth Extraction in the Posterior Maxilla: A Randomized, Split-Mouth, Controlled Trial.
Brief Title: The Effect of Alveolar Ridge Preservation After Tooth Extraction in the Posterior Maxilla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NYU College of Dentistry (Other)
Collaborators: Osteo Science Foundation (Unknown)
Responsible Party: Principal Investigator, Ismael Khouly, Associate Director of Periodontology & Implant Dentistry, NYU College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01597
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Tooth Extraction
Keywords: Alveolar Ridge Preservation; Xenograft bone graft; Collagen membrane
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Treatment (No Intervention): Tooth extraction with no bone graft.
- Alveolar Ridge Preservation Treatment (Active Comparator): Tooth extraction followed by alveolar ridge preservation using xenograft bone graft and covered by a resorbable collagen membrane.
  Interventions: Device: Xenograft

INTERVENTIONS:
Device: Xenograft
  Arms: Alveolar Ridge Preservation Treatment

SUMMARY:
This study is designed to assess the effects of Alveolar Ridge Preservation (ARP) after tooth extraction compared to extraction alone in the posterior maxilla. The results of this study will demonstrate if the use of ARP reduces alveolar ridge resorption at 6 months post extraction in the posterior maxilla region.

DETAILED DESCRIPTION:
Fifteen subjects requiring extraction of one posterior tooth in the right maxilla and one posterior tooth in the left maxilla will be considered for enrollment. Subjects who meet the inclusion and exclusion criteria will be randomized to receive alveolar ridge preservation on one side of the maxilla and only an extraction on the other side of the maxilla.

Extraction of the failing teeth will be performed atraumatically; a mucoperiosteal flap will not be employed. After removal of the tooth, the alveolus will be meticulously debrided and cleaned. In the test site, the socket will be filled with xenograft and a collagen membrane. In the control site, no graft material or collagen membrane will be used. Clinical measurements, standardized peri-apical radiographs and Cone Beam Computed Tomography scans will be performed immediately following tooth extractions (visit 2) and 6 months (visit 4) after extractions.

Subjects will be examined over the course of 6 months. Investigators will be trained prior to participating in the study. Training will be undertaken during a site initiation visit and will include a detailed description of all study procedures including treatment methods, and measurement methods to obtain study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily sign the informed consent form.
2. Subjects must be male or female who are at least 20-70 years of age.
3. Subjects must be able and willing to follow study procedures and instructions.
4. Presence of one posterior tooth in the right maxilla and one posterior tooth in the left maxilla that require extraction (ADA tooth positions 2-4 and 13-15). The same type of tooth should be in booth side, either two molars or two premolars.
5. Teeth extractions of one posterior tooth in the right maxilla and one posterior tooth in the left maxilla must be completed successfully (ADA tooth positions 2-4 and 13-15).
6. If present, teeth adjacent to the teeth slated for extraction must be healthy. Healthy teeth are defined as asymptomatic teeth without periapical lesions.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating, or who intend to become pregnant during the study period following entrance into the study.
2. Subjects who have failed to maintain good plaque control.
3. Subjects with any systemic condition such as uncontrolled diabetes mellitus, cancer, HIV, disorders that compromise wound healing, chronic high dose steroid therapy, intravenous and oral bisphosphonate therapy, bone metabolic diseases, history of irradiation of the head and neck area, or any other immuno-suppressive therapy that would contraindicate oral surgical treatment.
4. Subjects who report allergy or hypersensitivity to any of the products (collagen membrane and ABBM) used throughout the study.
5. Presence of ≥3 mm of vertical loss of the buccal bone in relation to the palatal wall.
6. Subjects with untreated periodontitis.
7. Presence of acute dentoalveolar infections in the teeth slated for extraction.
8. Subjects who are heavy smokers (defined as >10 cigarettes per day or >1 cigar per day) or chew tobacco, including within 3 months prior to enrollment.
9. Subjects with conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non- compliance or unreliability

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-09-27 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the bucco-palatal width of the alveolar ridge measured in mm. | 6 Months
  Changes in the bucco-palatal width of alveolar ridge from baseline to 6 months, measured using CBCT data.
Changes in the vertical height of the alveolar ridge measured in mm. | 6 Months
  Changes in the vertical height of the alveolar ridge measured using Cone Beam Computed Tomography (CBCT) data and periapical radiographs.

SECONDARY OUTCOMES:
Alveolar bone volumetric changes measured in mm. | 6 Months
  Alveolar bone volumetric changes measured using CBCT data and from dental impressions.
Changes in the distance from the alveolar crestal bone to the sinus floor measured in mm. | 6 months
  Changes in the distance from the alveolar crestal bone to the sinus floor using CBCT data and standardized periapical radiographs.
Bone density changes from measured in mm. | 6 Months
  Bone density changes measured using CBCT data.
Changes in keratinized mucosa width and thickness measured in mm. | 6 months
  Changes in keratinized mucosa width and thickness.
Correlation of soft tissue and buccal bone wall thickness measured in mm. | 6 months
  Correlation of soft tissue and buccal bone wall thickness on radiographic outcomes.
Subject satisfaction will be assessed through questionnaire. | 6 Months
  Subject satisfaction will be assessed using a Visual Analogue Scale (VAS) (scored from 0-100) after extraction (visit 2), at 2 weeks (visit 3) and 6 months (visit 4) following tooth extractions.
Need for additional bone augmentation, including sinus bone augmentation measured in mm. | 1.5 Years
  Need for additional bone augmentation, including sinus bone augmentation, prior to implant placement at 6 months post extractions
Implant success rate measured by percentage. | 6 Months
  Evaluate dental implant success, in case the subject receives dental implant following healing of alveolar ridge after teeth extractions

CONTACTS AND LOCATIONS:
Overall Officials: Ismael E. Khouly, DDS, MS, PhD, Principal Investigator — Bluestone Center for Clinical Research
Locations (1):
- Bluestone Center for Clinical Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo MG, Liljenberg B, Lindhe J. Dynamics of Bio-Oss Collagen incorporation in fresh extraction wounds: an experimental study in the dog. Clin Oral Implants Res. 2010 Jan;21(1):55-64. doi: 10.1111/j.1600-0501.2009.01854.x. PMID 20070748
- [Background] Araujo MG, Lindhe J. Socket grafting with the use of autologous bone: an experimental study in the dog. Clin Oral Implants Res. 2011 Jan;22(1):9-13. doi: 10.1111/j.1600-0501.2010.01937.x. Epub 2010 Nov 22. PMID 21091539
- [Background] Carmagnola D, Adriaens P, Berglundh T. Healing of human extraction sockets filled with Bio-Oss. Clin Oral Implants Res. 2003 Apr;14(2):137-43. doi: 10.1034/j.1600-0501.2003.140201.x. PMID 12656871
- [Background] Ashman A. Postextraction ridge preservation using a synthetic alloplast. Implant Dent. 2000;9(2):168-76. doi: 10.1097/00008505-200009020-00011. PMID 11307396
- [Background] Atieh MA, Alsabeeha NH, Payne AG, Duncan W, Faggion CM, Esposito M. Interventions for replacing missing teeth: alveolar ridge preservation techniques for dental implant site development. Cochrane Database Syst Rev. 2015 May 28;2015(5):CD010176. doi: 10.1002/14651858.CD010176.pub2. PMID 26020735
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Camargo PM, Lekovic V, Weinlaender M, Klokkevold PR, Kenney EB, Dimitrijevic B, Nedic M, Jancovic S, Orsini M. Influence of bioactive glass on changes in alveolar process dimensions after exodontia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Nov;90(5):581-6. doi: 10.1067/moe.2000.110035. PMID 11077380
- [Background] Greenstein G, Jaffin RA, Hilsen KL, Berman CL. Repair of anterior gingival deformity with durapatite. A case report. J Periodontol. 1985 Apr;56(4):200-3. doi: 10.1902/jop.1985.56.4.200. PMID 2987474
- [Background] Norton MR, Wilson J. Dental implants placed in extraction sites implanted with bioactive glass: human histology and clinical outcome. Int J Oral Maxillofac Implants. 2002 Mar-Apr;17(2):249-57. PMID 11958408
- [Background] Rasperini G, Canullo L, Dellavia C, Pellegrini G, Simion M. Socket grafting in the posterior maxilla reduces the need for sinus augmentation. Int J Periodontics Restorative Dent. 2010 Jun;30(3):265-73. PMID 20386783
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Soehren SE, Van Swol RL. The healing extraction site: a donor area for periodontal grafting material. J Periodontol. 1979 Mar;50(3):128-33. doi: 10.1902/jop.1979.50.3.128. PMID 285263